CLINICAL TRIAL: NCT00950404
Title: An Open-Label, Crossover Study In Healthy Volunteers To Evaluate The Pharmacokinetics Of Sildenafil Following Administration Of Three Orally Disintegrating Tablet Formulations Of Sildenafil Without Water Relative To Viagra Conventional Oral Tablet With Water.
Brief Title: Bioavailability of 3 Sildenafil Oral Disintegrating Tablet Formulations Compared to the Standard Oral Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A1481273
Record Dates: First submitted 2009-07-30; First posted 2009-07-31 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Healthy Volunteers
Keywords: Bioavailability Pharmacokinetic Formulation
MeSH Terms: interventions — Sildenafil Citrate; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Viagra 50 mg tablet, administered with water. (Active Comparator)
  Interventions: Drug: Viagra 50 mg tablet
- Formulation B ODT tablet 50 mg, administered without water. (Experimental)
  Interventions: Drug: Formulation B ODT tablet 50 mg
- Formulation C ODT tablet 50 mg, administered without water. (Experimental)
  Interventions: Drug: Formulation C ODT tablet 50 mg
- Formulation D ODT tablet 50 mg, administered without water. (Experimental)
  Interventions: Drug: Formulation D ODT tablet 50 mg

INTERVENTIONS:
Drug: Viagra 50 mg tablet — Commercial tablet, 50 mg, single dose administered with water
  Arms: Viagra 50 mg tablet, administered with water.
Drug: Formulation B ODT tablet 50 mg — Oral disintegrating tablet (ODT), 50 mg, single dose administered without water
  Arms: Formulation B ODT tablet 50 mg, administered without water.
Drug: Formulation C ODT tablet 50 mg — ODT, 50 mg, single dose administered without water
  Arms: Formulation C ODT tablet 50 mg, administered without water.
Drug: Formulation D ODT tablet 50 mg — ODT, 50 mg, single dose, administered without water
  Arms: Formulation D ODT tablet 50 mg, administered without water.

SUMMARY:
The bioavailability of the oral disintegrating tablet formulations given without water will be similar to an equivalent dose of the standard oral tablet given with water.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Weight: BMI from 17.5 to 30.5

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* A positive urine drug screen.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2009-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
AUC0-T and Cmax of sildenafil | 1 month

SECONDARY OUTCOMES:
AUC0-Tmax and AUCinf of sildenafil | 1 month
Tmax and half-life of sildenafil | 1 month
adverse events | 3 weeks
vital signs | 3 weeks
laboratory parameters | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481273&StudyName=Bioavailability%20of%203%20sildenafil%20oral%20disintegrating%20tablet%20formulations%20compared%20to%20the%20standard%20oral%20tablet